CLINICAL TRIAL: NCT00596050
Title: Ketamine Versus Etomidate for Procedural Sedation for Pediatric Orthopedic Reductions
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Drexel University College of Medicine (Other)
Responsible Party: Sponsor
Organization: Drexel University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 16271; Project No 1041266 (Other: drexel); Action No 47488 (Other: drexel); Detail No 240976 (Other: drexel)
Record Dates: First submitted 2008-01-07; First posted 2008-01-16 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Conscious Sedation Failure During Procedure
Keywords: procedural sedation; fracture reduction; pediatric emergency medicine; etomidate; ketamine; analgesia
MeSH Terms: conditions — Agnosia | interventions — Ketamine; Midazolam; Etomidate; Fentanyl; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ketamine and midazolam (Active Comparator): ketamine and midazolam
  Interventions: Drug: ketamine and midazolam
- etomidate and fentanyl and lidocaine (Active Comparator): etomidate and fentanyl and lidocaine
  Interventions: Drug: etomidate, fentanyl, and lidocaine

INTERVENTIONS:
Drug: ketamine and midazolam — ketamine 1 mg/kg/dose, midazolam 0.05 mg/kg/dose max 2 mg
  Arms: ketamine and midazolam
Drug: etomidate, fentanyl, and lidocaine — etomidate 0.2 mg/kg/dose, fentanyl 1 microgram/kg/dose, lidocaine 0.5 mg/kg/dose
  Arms: etomidate and fentanyl and lidocaine

SUMMARY:
There are multiple retrospective studies detailing the use of etomidate in pediatric procedural sedation but few to no prospective clinical trials. None have compared etomidate to ketamine, currently the most commonly used sedative in the emergency department for pediatric procedural sedation. The investigators propose a randomized, controlled trial comparing etomidate versus ketamine for procedural sedation for fracture reduction for children presenting with extremity fracture requiring sedation for reduction. The investigators hypothesize that etomidate in combination with fentanyl will have similar reduction of distress and procedural recall as ketamine in combination with midazolam.

DETAILED DESCRIPTION:
There are multiple retrospective studies detailing the use of etomidate in pediatric procedural sedation but few to no prospective clinical trials. None have compared etomidate to ketamine, currently the most commonly used sedative in the emergency department for pediatric procedural sedation. The investigators propose a randomized, controlled trial comparing etomidate versus ketamine for procedural sedation for fracture reduction for children presenting with extremity fracture requiring sedation for reduction. The investigators hypothesize that etomidate in combination with fentanyl will have similar reduction of distress and procedural recall as ketamine in combination with midazolam.

ELIGIBILITY:
Inclusion Criteria:

* age 5-18 years
* extremity fracture requiring reduction with sedation in emergency department

Exclusion Criteria:

* allergy to etomidate, midazolam, fentanyl, ketamine, lidocaine
* multi-system trauma
* history of psychosis
* pregnancy
* illicit drug use
* developmental delay
* non-english speaker

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2006-08; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
OSBD-r | immediate
  Outcome measures included guardian and staff completion of visual analog scale and Likert scales for observed pain and satisfaction, blinded OSBD-r (Observational Scale of Behavioral Distress-Revised) scoring of digital recordings of reductions, and sedation and recovery times.

SECONDARY OUTCOMES:
Likert satisfaction scale | immediate
  Outcome measures included guardian and staff completion of visual analog scale and Likert scales for observed pain and satisfaction, blinded OSBD-r (Observational Scale of Behavioral Distress-Revised) scoring of digital recordings of reductions, and sedation and recovery times.
procedural recall | immediate
  Outcome measures included guardian and staff completion of visual analog scale and Likert scales for observed pain and satisfaction, blinded OSBD-r (Observational Scale of Behavioral Distress-Revised) scoring of digital recordings of reductions, and sedation and recovery times.

CONTACTS AND LOCATIONS:
Overall Officials: Jannet J Lee-Jayaram, M.D., Principal Investigator — Drexel University College of Medicine
Locations (1):
- St. Christopher's Hospital for Children, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bahn EL, Holt KR. Procedural sedation and analgesia: a review and new concepts. Emerg Med Clin North Am. 2005 May;23(2):503-17. doi: 10.1016/j.emc.2004.12.013. PMID 15829394
- [Background] Kennedy RM, Porter FL, Miller JP, Jaffe DM. Comparison of fentanyl/midazolam with ketamine/midazolam for pediatric orthopedic emergencies. Pediatrics. 1998 Oct;102(4 Pt 1):956-63. doi: 10.1542/peds.102.4.956. PMID 9755272
- [Background] Acworth JP, Purdie D, Clark RC. Intravenous ketamine plus midazolam is superior to intranasal midazolam for emergency paediatric procedural sedation. Emerg Med J. 2001 Jan;18(1):39-45. doi: 10.1136/emj.18.1.39. PMID 11310461
- [Background] Gerardi MJ, Sacchetti AD, Cantor RM, Santamaria JP, Gausche M, Lucid W, Foltin GL. Rapid-sequence intubation of the pediatric patient. Pediatric Emergency Medicine Committee of the American College of Emergency Physicians. Ann Emerg Med. 1996 Jul;28(1):55-74. doi: 10.1016/s0196-0644(96)70140-3. PMID 8669740
- [Background] Ruth WJ, Burton JH, Bock AJ. Intravenous etomidate for procedural sedation in emergency department patients. Acad Emerg Med. 2001 Jan;8(1):13-8. doi: 10.1111/j.1553-2712.2001.tb00539.x. PMID 11136141
- [Background] Vinson DR, Bradbury DR. Etomidate for procedural sedation in emergency medicine. Ann Emerg Med. 2002 Jun;39(6):592-8. doi: 10.1067/mem.2002.123695. PMID 12023700
- [Background] Dickinson R, Singer AJ, Carrion W. Etomidate for pediatric sedation prior to fracture reduction. Acad Emerg Med. 2001 Jan;8(1):74-7. doi: 10.1111/j.1553-2712.2001.tb00558.x. PMID 11136155
- [Background] Schenarts CL, Burton JH, Riker RR. Adrenocortical dysfunction following etomidate induction in emergency department patients. Acad Emerg Med. 2001 Jan;8(1):1-7. doi: 10.1111/j.1553-2712.2001.tb00537.x. PMID 11136139
- [Background] Godambe SA, Elliot V, Matheny D, Pershad J. Comparison of propofol/fentanyl versus ketamine/midazolam for brief orthopedic procedural sedation in a pediatric emergency department. Pediatrics. 2003 Jul;112(1 Pt 1):116-23. doi: 10.1542/peds.112.1.116. PMID 12837876
- [Background] Scott J, Huskisson EC. Graphic representation of pain. Pain. 1976 Jun;2(2):175-84. No abstract available. PMID 1026900
- [Background] Keim SM, Erstad BL, Sakles JC, Davis V. Etomidate for procedural sedation in the emergency department. Pharmacotherapy. 2002 May;22(5):586-92. doi: 10.1592/phco.22.8.586.33204. PMID 12013357
- [Background] Mace SE, Barata IA, Cravero JP, Dalsey WC, Godwin SA, Kennedy RM, Malley KC, Moss RL, Sacchetti AD, Warden CR, Wears RL; American College of Emergency Physicians. Clinical policy: evidence-based approach to pharmacologic agents used in pediatric sedation and analgesia in the emergency department. Ann Emerg Med. 2004 Oct;44(4):342-77. doi: 10.1016/j.annemergmed.2004.04.012. No abstract available. PMID 15459618
- [Background] Jay SM, Ozolins M, Elliott C, Caldwell S. Assessment of children's distress during painful medical procedures. J Health Psycho. 1983; 2: 133-147